CLINICAL TRIAL: NCT02188121
Title: Fixed Dose Intervention Trial of New England Enhancing Survival in Serious Mental Illness Patients
Brief Title: Fixed Dose Intervention Trial of New England Enhancing Survival in SMI Patients
Acronym: FITNESS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Michael J. Gill Mental Health Clinic (Other); Massachusetts Mental Health Center (Other); Dauten Family Center for Bipolar Treatment Innovation at Massachusetts General Hospital (Unknown); The Edinburg Center (Other)
Responsible Party: Principal Investigator, Dost Ongur, Chief of Psychotic Disorders Division at McLean Hospital and Associate Professor in Psychiatry at Harvard Medical School, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014P001599
Record Dates: First submitted 2014-07-08; First posted 2014-07-11 (Estimated); Results first posted 2022-11-22 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Serious Mental Illness; Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Cardiovascular Disease; Major Depressive Disorder; Psychosis NOS
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Cardiovascular Diseases; Depressive Disorder, Major; Mental Disorders | interventions — Simvastatin; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Statin and/or Angiotensin Receptor Blocker (Experimental): Simvastatin 20mg PO daily and/or Losartan 25mg PO daily
  Interventions: Drug: Simvastatin; Drug: Losartan
- Usual treatment (No Intervention): We will compare the initial treatment intervention with usual treatment (control arm), with both arms superimposed on a system of regular monitoring base. The investigators will make no effort to alter or influence treatment or use of that treatment for subjects in the control arm. Note that our goal in the Control arm is to characterize "usual treatment". We will not intervene in this care except in emergencies. Some patients who need care for metabolic syndrome may not be receiving it - just as they would if not in our trial.

INTERVENTIONS:
Drug: Simvastatin — 3-hydroxy-3-methylglutaryl-coenzyme (HMG-CoA) reductase inhibitors
  Arms: Statin and/or Angiotensin Receptor Blocker
Drug: Losartan — Angiotensin II receptor antagonist
  Arms: Statin and/or Angiotensin Receptor Blocker

SUMMARY:
Patients with severe mental illness (SMI) die younger than persons in the general population. Much of the excess mortality for SMI patients is attributable to cardiovascular disease, and is exacerbated by treatment with second-generation antipsychotics (2GAs). Although the cardiovascular risks are well-known, and safe, efficacious therapy exists, few SMI patients receive cardiovascular prevention drugs. Care delivery fragmentation and poor patient adherence are central problems to reducing cardiovascular risks for patients with SMI. To address these problems, we propose to conduct a multi-site, open-label, randomized controlled trial comparing an initial treatment strategy of free, fixed-doses of two generic, cardiovascular prevention drugs (statins and angiotensin drugs) delivered within mental health clinics versus usual treatment. The study will include adult patients (18+ years old) with schizophrenia, schizoaffective disorder, bipolar disorder, major depressive disorder, or psychosis not otherwise specified (NOS) who have received 2GAs treatment within the past six months from within four mental health clinics in the Boston area. We have three aims: 1) to compare the proportions of subjects in each arm who are receiving cardiovascular drug treatment and are adherent to therapy during 12-months of follow-up; 2) to compare changes in composite (e.g., Framingham scores) and individual (e.g., lipid levels) cardiovascular risk factor levels using an intent-to-treat (ITT) approach; and 3) to compare risk factor levels, accounting for variation in adherence over time, using causal inference techniques to estimate the per-protocol effect of the intervention. Our three aims examine whether this low cost, streamlined treatment strategy increases the numbers of subjects receiving cardiovascular prevention therapy and improves cardiovascular risk levels. We will follow subjects for 12 months, and collect interview and biometric data at baseline and over the following 12 months. Subjects will have the option to continue for another 12 months, during which we will continue to collect interview and biometric data, but will not prescribe cardiovascular medications. This population-based initial treatment strategy could be an effective and efficient approach for overcoming traditional barriers to cardiovascular disease prevention within the SMI population. Findings from this study will inform efforts to improve care and outcomes, and to enhance survival for patients with severe mental illness.

DETAILED DESCRIPTION:
By design, all subjects in the Intervention arm will start by being under treatment. During the course of follow-up, we expect that some will stay consistently on treatment, some will discontinue treatment (become non-adherent), while others will make transitions on and off treatment in various patterns. In contrast, by design, subjects in the Usual Treatment (control) arm do not start on treatment; however, some will initiate treatment as a result of usual clinical care, e.g., primary care physician initiation. At any point we will be comparing two binary outcomes (on or off treatment) and will use standard methods for comparing two proportions to test statistical significance and get confidence intervals for the difference in the percent on treatment in the two arms. Participants who are ineligible for randomization will be followed similarly to participants in the Usual Treatment Arm, in a third, non-randomized group, which will be excluded from the primary analysis.

ELIGIBILITY:
Inclusion Criteria:

* Incident or prevalent cases: schizophrenia, schizoaffective disorder, bipolar disorder, major depressive disorder, or psychosis NOS (chart diagnosis).
* Age 18 years and older.
* Recent treatment with a standing 2GA, e.g., receiving a standing 2GA in the past 6 months.
* Concomitant psychotropic medications will be allowed.
* Ongoing treatment of their mental illnesses at one of four study mental health clinics, defined as entering one of the two-year First Episode Clinic treatment programs as a de novo patient (new disease) or having been diagnosed >2 years ago and had at least six visits in the past 12 months (prevalent disease).

Exclusion Criteria:

* • Unstable/active disease or potential contraindications with both study medications, e.g., diabetes, unstable angina or recent acute coronary syndrome, pregnancy, very high risk factors on the screening labs (e.g., A1c>7%), renal failure, liver failure, or both statin and angiotension drug contraindications.

  * Unable to provide informed consent, e.g., has dementia, developmental disability, other cognitive disorder, or fails screening mini-mental status exam (subjects with guardians may participate with guardian consent)
  * Receiving active cardiovascular treatment, defined as receiving both a statin or ARB in the past three months.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2015-02; Primary Completion 2020-10 (Actual); Study Completion 2021-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dost Ongur, MD PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

REFERENCES:
- [Derived] Chouinard VA, Price M, Forte S, Prete S, Heinrich H, Smith SN, Fung V, Hsu J, Ongur D. Baseline Cardiovascular Risk Factors in Patients With Severe Mental Illness (SMI) and Second Generation Antipsychotic Use From the Fixed Dose Intervention Trial of New England Enhancing Survival in SMI (FITNESS). J Clin Psychiatry. 2025 Jan 8;86(1):24m15392. doi: 10.4088/JCP.24m15392. PMID 39832344

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 23 participants were excluded after enrollment but prior to assignment to a study arm. The reasons for exclusion were vital signs or lab values outside of inclusion criteria, or emergence of details after enrollment that made participant ineligible.
Period: Overall Study
Arm/Group | Statin and/or Angiotensin Receptor Blocker | Usual Treatment
Started | 99 | 105
Completed | 79 | 78
Not Completed | 20 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Statin and/or Angiotensin Receptor Blocker | Usual Treatment | Total
Number analyzed (Participants) | 99 | 105 | 204
Age, Continuous [Mean (Full Range); unit: years] | 36.0 [18 to 68] | 38.3 [19 to 74] | 37.2 [18 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 46 | 81
  Male | 64 | 59 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 5 | 15
  Not Hispanic or Latino | 85 | 92 | 177
  Unknown or Not Reported | 4 | 8 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 19 | 34
  White | 70 | 75 | 145
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 8 | 4 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 99 | 105 | 204

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants on Adequate Cardiovascular Prevention Care (Defined as Taking a Statin and Angiotensin Medication)
Time Frame: Baseline to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Statin and/or Angiotensin Receptor Blocker | Usual Treatment
Number analyzed (Participants) | 99 | 105
Participants | 66 | 8

2. Secondary Outcome: Change in Low Density Lipoprotein Levels
Description: Similar to secondary outcome measure but focusing on Low Density Lipoprotein, Systolic Blood Pressure, and Hemoglobin A1c
Time Frame: Baseline to 12 months
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Statin and/or Angiotensin Receptor Blocker | Usual Treatment
Number analyzed (Participants) | 99 | 105
mg/dL
  Baseline | 100 [96 to 105] | 106 [101 to 117]
  12 months | 86 [82 to 96] | 100 [97 to 117]

3. Other Pre Specified Outcome: Change in Modified Framingham Score as a Summary Cardiovascular Risk Level
Description: The outcome here is the difference in summary risk level changes (e.g., modified Framingham score) between our two study groups, i.e., do intervention subjects experience differential changes in cardiovascular risk levels compared to control subjects. This outcome will be continuously measured (but not necessarily normally distributed).
Time Frame: Baseline and 3, 6, 9, and 12 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change in Number of Distinct Cardiovascular Prevention Drugs Taken
Description: Similar to primary outcome measure, but here we count the number of distinct cardiovascular prevention drugs taken by the patient as a continuous measure to reflect potential for partial treatment.
Time Frame: Baseline and 3, 6, 9, and 12 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Systolic Blood Pressure
Description: Similar to secondary outcome measure but focusing on Systolic Blood Pressure
Time Frame: Baseline and 3, 6, 9, and 12 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Hemoglobin A1C
Description: Similar to secondary outcome measure but focusing on Hemoglobin A1c
Time Frame: Baseline and 3, 6, 9, and 12 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Percent on Adequate Cardiovascular Prevention Care
Time Frame: Baseline to 3 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Percent on Adequate Cardiovascular Prevention Care
Time Frame: Baseline to 6 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Percent on Adequate Cardiovascular Prevention Care
Time Frame: Baseline to 9 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Mean Percentage of Follow up Time During Which Each Group is on Adequate Cardiovascular Prevention Care
Time Frame: Baseline to 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years per participant
Arm/Group | Statin and/or Angiotensin Receptor Blocker | Usual Treatment
All-Cause Mortality (participants affected / at risk) | 1/99 | 2/105
Serious Adverse Events (participants affected / at risk) | 7/99 | 4/105
Other Adverse Events (participants affected / at risk) | 72/99 | 50/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Statin and/or Angiotensin Receptor Blocker (N=99) | Usual Treatment (N=105)
Elevated creatine kinase level (Blood and lymphatic system disorders) | 2 | 0 — Classified as severe if >2x normal range
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypotension (Cardiac disorders) | 1 | 0
Dehydration (General disorders) | 1 | 0
Leukemia (Blood and lymphatic system disorders) | 1 | 0
Placed on Lithium while on Losartan (General disorders) | 1 | 0 — This is a relative contraindication. Patient taken off of losartan when team informed going on lithium. No sequelae
Diabetes (Endocrine disorders) | 0 | 1 — New onset
Suicide attempt (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Statin and/or Angiotensin Receptor Blocker (N=99) | Usual Treatment (N=105)
Psychiatric Hospitalization (Psychiatric disorders) | 23 | 20
Medical Hospitalization (General disorders) | 6 | 7
Laboratory values outside normal range (General disorders) | 43 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/21/NCT02188121/Prot_002.pdf
  • Statistical Analysis Plan (2018-02-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT02188121/SAP_001.pdf